CLINICAL TRIAL: NCT01025375
Title: Effects of Inulin on Satiety and Food Intake
Acronym: Inulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: HumBio_Westerterp08_2
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Obesity
Keywords: overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Inulin; oligofructose; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: inulin — 10gram/day inulin for 13-day treatment
  Other Names: oligofructose
Dietary Supplement: inulin — 16gram/day inulin for 13-day treatment
  Other Names: oligofructose
Dietary Supplement: placebo — 16gram/day maltodextrin (placebo) for 13-day treatment
  Other Names: maltodextrin

SUMMARY:
To assess the effect of inulin on appetite profile ratings, food intake and satiety hormones.

DETAILED DESCRIPTION:
Based upon a slower digestion and the fermentation in the intestinal tract, food containing soluble dietary fibres, such as inulin, is hypothesized to be more satiating, and to limit energy intake, in humans. Does supplementation of inulin (at 2 dosages) versus placebo over 13 consecutive days in normal to overweight men and women, lead to an increase in satiety, a reduction in food intake and stronger postprandial increases in GLP-1 and PYY?

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 60 years
* BMI between 23 and 28 kg/m2
* dietary unrestraint (TFEQ: F1<9)

Exclusion Criteria:

* age under 18 and above 60 years
* BMI under 23 and above 28 kg/m2
* dietary restraint (TFEQ: F1>9)
* use of medication
* pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
food intake | on testday 0 and 13

SECONDARY OUTCOMES:
appetite profile ratings | on test day 0, 8 and 13 (at 16 time points)
satiety hormones (GLP-1 and PYY) | on test day 0 and 13 (at 9 time points

CONTACTS AND LOCATIONS:
Overall Officials: Klaas R Westerterp, Prof, Principal Investigator — NUTRIM
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands